CLINICAL TRIAL: NCT00875069
Title: Efficacy and Safety of Ethanol Lock Solution in Prevention of Catheter Related Bloodstream Infection for Patients Suffering Acute Renal Failure, and Hospitalized in Intensive Care Unit. A Multi-Center, Randomized, Versus Placebo, Double Blinded Clinical Trial.
Acronym: ELVIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHU-0050
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Acute Renal Failure; Infection
Keywords: Nosocomial infection; Catheterization; Central Venous Ethanol; lock solution; intensive care units; Renal replacement therapy in ICU
MeSH Terms: conditions — Acute Kidney Injury; Infections; Cross Infection | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ethanol (Experimental)
  Interventions: Other: Ethanol
- placebo (Placebo Comparator)
  Interventions: Other: Ethanol

INTERVENTIONS:
Other: Ethanol — Dialysis catheter lock performed after renal replacement therapy session. Lock is instilling ethanol (or placebo) in each catheter lumen for 2 minutes before being withdrawn.

SUMMARY:
The primary objective of the study is to demonstrate the efficacy of 60% ethanol lock solution in preventing major catheter related infections in critically ill patients.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate the efficacy of 60% ethanol lock solution in preventing major catheter related infections in critically ill patients

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, over 18 years,
* Patients admitted in ICU
* Dialysis catheter insertion for renal replacement therapy
* At least two renal replacement therapy sessions
* Written informed consent
* Social security

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient requiring dialysis on arteriovenous fistula or permanent catheter
* Known allergy to ethanol
* Dialysis catheter covered or impregnated with antimicrobial agent
* Dialysis catheter insertion before ICU admission
* Single-lumen dialysis catheters
* Patient whose death is likely to occur within hours after admission to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1460 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The number of major catheter-related infections (CRI) defined as either catheter-related clinical sepsis without bloodstream infection or catheter-related bloodstream infection (CRBSI), during the ICU stay | after renal replacement therapy session

SECONDARY OUTCOMES:
frequencies of catheter colonization, severe mechanical complications, and adverse events | for two minutes before being withdrawn

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Souweine, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Soum E, Timsit JF, Ruckly S, Gruson D, Canet E, Klouche K, Argaud L, Garrouste-Orgeas M, Mariat C, Vincent F, Cayot S, Darmon M, Bohe J, Schwebel C, Bouadma L, Dupuis C, Souweine B, Lautrette A. Predictive factors for severe long-term chronic kidney disease after acute kidney injury requiring renal replacement therapy in critically ill patients: an ancillary study of the ELVIS randomized controlled trial. Crit Care. 2022 Nov 29;26(1):367. doi: 10.1186/s13054-022-04233-4. PMID 36447221
- [Derived] Iachkine J, Buetti N, de Grooth HJ, Briant AR, Mimoz O, Megarbane B, Mira JP, Ruckly S, Souweine B, du Cheyron D, Mermel LA, Timsit JF, Parienti JJ. Development and validation of a multivariable prediction model of central venous catheter-tip colonization in a cohort of five randomized trials. Crit Care. 2022 Jul 7;26(1):205. doi: 10.1186/s13054-022-04078-x. PMID 35799302
- [Derived] Almeida BM, Moreno DH, Vasconcelos V, Cacione DG. Interventions for treating catheter-related bloodstream infections in people receiving maintenance haemodialysis. Cochrane Database Syst Rev. 2022 Apr 1;4(4):CD013554. doi: 10.1002/14651858.CD013554.pub2. PMID 35363884
- [Derived] Boyer A, Timsit JF, Klouche K, Canet E, Phan TN, Bohe J, Rubin S, Orieux A, Lautrette A, Gruson D, Souweine B. Aminoglycosides in Critically Ill Septic Patients With Acute Kidney Injury Receiving Continuous Renal Replacement Therapy: A Multicenter, Observational Study. Clin Ther. 2021 Jun;43(6):1116-1124. doi: 10.1016/j.clinthera.2021.04.011. Epub 2021 May 24. PMID 34039478
- [Derived] Souweine B, Lautrette A, Gruson D, Canet E, Klouche K, Argaud L, Bohe J, Garrouste-Orgeas M, Mariat C, Vincent F, Cayot S, Cointault O, Lepape A, Guelon D, Darmon M, Vesin A, Caillot N, Schwebel C, Boyer A, Azoulay E, Bouadma L, Timsit JF. Ethanol lock and risk of hemodialysis catheter infection in critically ill patients. A randomized controlled trial. Am J Respir Crit Care Med. 2015 May 1;191(9):1024-32. doi: 10.1164/rccm.201408-1431OC. PMID 25668557